CLINICAL TRIAL: NCT02819388
Title: Evaluation of a Counseling Intervention to Improve Contraceptive Use in Deprived Neighborhoods: SIRIAN Randomized Controlled Trial.
Brief Title: Evaluation of a Contraceptive Counseling Intervention in Deprived Neighborhoods: SIRIAN Randomized Controlled Trial
Acronym: SIRIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Elia Diez David, Head of the Service of Programs and Preventive Interventions. Barcelona Public Health Agency, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ediezSIRIAN
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Contraception
Keywords: randomized control trial; contraception; inequalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Contraceptive counseling
  Interventions: Behavioral: Contraceptive counseling
- Control (No Intervention): Control group without counseling

INTERVENTIONS:
Behavioral: Contraceptive counseling — A culturally adapted counselling session lasting up to 45 minutes at the community setting. The interview is based in WHO guidelines and communication tools, in social cognitive theory and in motivational interviewing. Along the interview, topics follow easy to read leaflets prepared to discuss the main benefits of contraception from the view of the immigrant communities, with guided discussions on family planning in the life course, the amount of time required to care children, the economic resources that newborn and children need, and an assessment of the knowledge on the contraceptive methods, and of their current use. Contraceptive methods, abortion and emergency contraception are discussed. Primary health care centre and sexual and reproductive health clinic access is reinforced.
  Arms: Intervention

SUMMARY:
This study evaluates the effects of a community-based counseling intervention to improve contraception among residents in two deprived neighborhoods in Barcelona (Spain). Half of the participants received contraceptive counseling at the community setting, while the other half acted as a control group.

DETAILED DESCRIPTION:
To evaluate the effects of a community-based counseling intervention to improve contraception among residents in deprived neighborhoods a randomized controlled trial is performed. Women aged 14-49 years and men aged 14-39 years from two low income neighborhoods in Barcelona (Catalonia, Spain) who had not undergone an irreversible contraceptive method and aren't planning a pregnancy have been recruited in 2011-13. The intervention consists of a culturally developed and theoretically-based brief counseling in community settings. The primary outcome is the consistent use of very effective contraceptive methods (optimal use). Secondary outcomes analyzed are the incorrect use of very effective contraceptive methods and use of less effective methods stratified by sex and migrant status. Differences within subgroups from baseline to 3 months - follow up are analyzed and intervention effects are assessed with adjusted robust Poisson regressions.

ELIGIBILITY:
Inclusion Criteria:

* Women living in the selected neighbourhoods aged 14-49 years
* Men living in the selected neighbourhoods aged 14-39 years

Exclusion Criteria:

* Having undergone an irreversible contraceptive method
* Whishing or planning a pregnancy in the next year

Ages: 14 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of participants using consistently effective contraceptive methods (optimal use) assessed by questionnaire | Three months after the baseline
  Primary outcome is the consistent use of effective methods. Effective methods include female sterilization, vasectomy, tube obstruction, IUD, implants, oral contraception, rings, patches, injections and female and male condoms

SECONDARY OUTCOMES:
Number of participants inconsistently using effective methods assessed by questionnaire | Three months after the baseline
  Inconsistent use of effective methods: Condoms used in some intercourse episodes and not others, condoms used improperly, taking birth control pills but missing too many doses for pregnancy prevention
Number of participants using less effective methods (withdrawal and periodic abstinence) assessed by questionnaire | Three months after the baseline
  Use of less effective methods (withdrawal and periodic abstinence). Practices such as douching are not considered a contraceptive method

CONTACTS AND LOCATIONS:
Overall Officials: Elia Diez, MD, Principal Investigator — Agència de Salut Pública de Barcelona - Barcelna Public Health Agency
Locations (1):
- Agència de Salut Pública de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided